CLINICAL TRIAL: NCT06339996
Title: To Investigate Supplements for Improving Male Sperm Quality and Combating Aging
Brief Title: Male Supplements for Sperm Quality and Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Doctor, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH24-CT1-10
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Unrecognized Condition
Keywords: Male supplement; Sperm quality; Aging; Mitochondrial function; Sexual function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Male dietary supplement (Experimental): Patients received male supplements for a three-month treatment period
  Interventions: Dietary Supplement: Male supplement

INTERVENTIONS:
Dietary Supplement: Male supplement — Participants will be administered supplements for a three-month treatment period

SUMMARY:
This study investigates the effects of a new supplement on sperm quality in men with poor sperm quality. Fifty patients will receive the supplement for three months, followed by semen analysis and assessment of sperm aging and mitochondrial function. Changes in sexual function and aging symptoms will also be evaluated.

DETAILED DESCRIPTION:
Due to modern lifestyle factors such as high work pressure, stressful routines, and environmental pollution, there has been a significant decline in sperm quality among men, potentially leading to infertility. In response, various supplements have emerged claiming to enhance sperm quality. This prospective investigation aims to determine the efficacy of a new supplement in improving sperm quality among patients with poor sperm quality. The study will enroll 50 patients undergoing semen analysis at our reproductive center, administering the supplement over a three-month treatment period to those identified with poor sperm quality. Subsequent semen analysis will be conducted, alongside assessments of sperm mitochondrial metabolic function before and after supplement administration. Sexual function and aging symptoms will also be evaluated using the International Index of Erectile Function (IIEF-5) and the Aging Males Symptoms Scale (AMS) before and after the supplementation period. The study aims to compare differences in semen analysis, sperm mitochondrial metabolic function, sexual function, and aging symptoms before and after supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Not meet the criteria of the 6th edition of the WHO manual for human semen analysis
* BMI:18-30 kg/m2

Exclusion Criteria:

* Azoospermia
* Varicocele
* Chromosome anomaly
* Malignancy
* Using hormone therapy or supplements in recent 3 months

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Semen analysis | through study completion, an average of 1 year
  semen concentration, motility and morphology

SECONDARY OUTCOMES:
oxygen consumption of mitochondria | through study completion, an average of 1 year
  oxygen consumption rate
mitochondrial function | through study completion, an average of 1 year
  adenosine triphosphate production
sexual function | through study completion, an average of 1 year
  International Index of Erectile Function (IIEF-5): a diagnostic tool for erectile dysfunction. The scores for the IIEF-5 range from 5 to 25. Higher scores mean a worse outcome
aging symptoms | through study completion, an average of 1 year
  Aging Males Symptoms Scale (AMS): a simple and effective way to detect whether you may have andropause. Each item is rated on a scale of 1 to 5. There are 17 in total, so the minimum score is 17 and the maximum score is 85. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal A, Baskaran S, Parekh N, Cho CL, Henkel R, Vij S, Arafa M, Panner Selvam MK, Shah R. Male infertility. Lancet. 2021 Jan 23;397(10271):319-333. doi: 10.1016/S0140-6736(20)32667-2. Epub 2020 Dec 10. PMID 33308486
- [Background] Eisenberg ML, Esteves SC, Lamb DJ, Hotaling JM, Giwercman A, Hwang K, Cheng YS. Male infertility. Nat Rev Dis Primers. 2023 Sep 14;9(1):49. doi: 10.1038/s41572-023-00459-w. PMID 37709866
- [Background] Wang C, Mbizvo M, Festin MP, Bjorndahl L, Toskin I; other Editorial Board Members of the WHO Laboratory Manual for the Examination and Processing of Human Semen. Evolution of the WHO "Semen" processing manual from the first (1980) to the sixth edition (2021). Fertil Steril. 2022 Feb;117(2):237-245. doi: 10.1016/j.fertnstert.2021.11.037. Epub 2022 Jan 5. PMID 34996596
- [Background] Hussein HA, Hassaneen ASA, Ali ME, Sindi RA, Ashour AM, Fahmy SM, Swelum AA, Ahmed AE. The Impact of Rumen-Protected L-Arginine Oral Supplementation on Libido, Semen Quality, Reproductive Organ Biometry, and Serum Biochemical Parameters of Rams. Front Vet Sci. 2022 Jun 24;9:899434. doi: 10.3389/fvets.2022.899434. eCollection 2022. PMID 35812886
- [Background] Shin D, Jeon SH, Piao J, Park HJ, Tian WJ, Moon DG, Ahn ST, Jeon KH, Zhu GQ, Park I, Park HJ, Bae WJ, Cho HJ, Hong SH, Kim SW. Efficacy and Safety of Maca (Lepidium meyenii) in Patients with Symptoms of Late-Onset Hypogonadism: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. World J Mens Health. 2023 Jul;41(3):692-700. doi: 10.5534/wjmh.220112. Epub 2023 Jan 1. PMID 36593713
- [Background] Lee HW, Lee MS, Qu F, Lee JW, Kim E. Maca (Lepidium meyenii Walp.) on semen quality parameters: A systematic review and meta-analysis. Front Pharmacol. 2022 Aug 30;13:934740. doi: 10.3389/fphar.2022.934740. eCollection 2022. PMID 36110519
- [Background] Brahmajosyula M, Morimoto Y. Exogenous GSH Supplementation to Raw Semen Alters Sperm Kinematic Parameters in Infertile Patients. Reprod Sci. 2023 Sep;30(9):2853-2865. doi: 10.1007/s43032-023-01221-z. Epub 2023 Apr 3. PMID 37012490
- [Background] Alahmar AT. Coenzyme Q10 improves sperm motility and antioxidant status in infertile men with idiopathic oligoasthenospermia. Clin Exp Reprod Med. 2022 Dec;49(4):277-284. doi: 10.5653/cerm.2022.05463. Epub 2022 Nov 4. PMID 36482502
- [Background] Nadjarzadeh A, Shidfar F, Amirjannati N, Vafa MR, Motevalian SA, Gohari MR, Nazeri Kakhki SA, Akhondi MM, Sadeghi MR. Effect of Coenzyme Q10 supplementation on antioxidant enzymes activity and oxidative stress of seminal plasma: a double-blind randomised clinical trial. Andrologia. 2014 Mar;46(2):177-83. doi: 10.1111/and.12062. Epub 2013 Jan 7. PMID 23289958
- [Background] Wang R, Wang S, Song Y, Zhou H, Pan Y, Liu L, Niu S, Liu X. Effect of vitamin E on Semen Quality Parameters: A Meta-Analysis of a Randomized Controlled Trial. Urol J. 2022 Nov 8;19(5):343-351. doi: 10.22037/uj.v19i.7160. PMID 36029025
- [Background] Alahmar AT. The Effect of Selenium Therapy on Semen Parameters, Antioxidant Capacity, and Sperm DNA Fragmentation in Men with Idiopathic Oligoasthenoteratospermia. Biol Trace Elem Res. 2023 Dec;201(12):5671-5676. doi: 10.1007/s12011-023-03638-8. Epub 2023 Mar 23. PMID 36959435
- [Background] Schisterman EF, Sjaarda LA, Clemons T, Carrell DT, Perkins NJ, Johnstone E, Lamb D, Chaney K, Van Voorhis BJ, Ryan G, Summers K, Hotaling J, Robins J, Mills JL, Mendola P, Chen Z, DeVilbiss EA, Peterson CM, Mumford SL. Effect of Folic Acid and Zinc Supplementation in Men on Semen Quality and Live Birth Among Couples Undergoing Infertility Treatment: A Randomized Clinical Trial. JAMA. 2020 Jan 7;323(1):35-48. doi: 10.1001/jama.2019.18714. PMID 31910279
- [Background] Irani M, Amirian M, Sadeghi R, Lez JL, Latifnejad Roudsari R. The Effect of Folate and Folate Plus Zinc Supplementation on Endocrine Parameters and Sperm Characteristics in Sub-Fertile Men: A Systematic Review and Meta-Analysis. Urol J. 2017 Aug 29;14(5):4069-4078. PMID 28853101
- [Background] Zhao J, Dong X, Hu X, Long Z, Wang L, Liu Q, Sun B, Wang Q, Wu Q, Li L. Zinc levels in seminal plasma and their correlation with male infertility: A systematic review and meta-analysis. Sci Rep. 2016 Mar 2;6:22386. doi: 10.1038/srep22386. PMID 26932683
- [Background] Taravati A, Tohidi F. Association between seminal plasma zinc level and asthenozoospermia: a meta-analysis study. Andrologia. 2016 Aug;48(6):646-53. doi: 10.1111/and.12494. Epub 2015 Nov 5. PMID 26541500
- [Background] Dimitriadis F, Borgmann H, Struck JP, Salem J, Kuru TH. Antioxidant Supplementation on Male Fertility-A Systematic Review. Antioxidants (Basel). 2023 Mar 30;12(4):836. doi: 10.3390/antiox12040836. PMID 37107211
- [Background] Li KP, Yang XS, Wu T. The Effect of Antioxidants on Sperm Quality Parameters and Pregnancy Rates for Idiopathic Male Infertility: A Network Meta-Analysis of Randomized Controlled Trials. Front Endocrinol (Lausanne). 2022 Feb 21;13:810242. doi: 10.3389/fendo.2022.810242. eCollection 2022. PMID 35265037